CLINICAL TRIAL: NCT03770585
Title: Comparative Study Between Fluoroscopy Guided Lumbar Facet Joint Injection Versus Ultrasound Guided Injection in Patients With Low Back Pain Due to Facet Syndrome
Brief Title: Fluoroscopy Guided Lumbar Facet Joint Injection Versus Ultrasound Guided Injection in Patients With Low Back Pain Due to Facet Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Collaborators: Tanta University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 30476/08/15
Record Dates: First submitted 2017-03-25; First posted 2018-12-10 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Facet Syndrome of Lumbar Spine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1(Fluoroscopy guided group) (Active Comparator): IN Fluoroscopy guided group, with x-ray beam, after cleaning and drapping and administration of local anesthesia, a22-g spinal needle is inserted in line till bony contact is felt under sterile conditions. Each facet joint is infiltrated with a mixture containing 0.5 ml of 0.25 % bupivacaine and 0.5 ml (20mg) methylprednisolone acetate injected into the joint.
  Interventions: Procedure: Fluoroscopy guided Facet joint injection
- Group2 (Ultrasound guided group) (Active Comparator): In Ultrasound guided group, with Ultrasound guidance, , a mixture containing 0.5 ml of 0.25 % bupivacaine and 0.5 ml(20mg) methylprednisolone acetate is administered intra-articular (until resistance was encountered) and injected around the posterior facet joint capsule.
  Interventions: Procedure: Ultrsound guided Facet joint injection

INTERVENTIONS:
Procedure: Fluoroscopy guided Facet joint injection — Fluoroscopy guided Facet joint injection (The patient will be placed in the prone position with a pillow under the abdomen to correct the lumbar lordosis. The joint to be injected is located and marked, the x ray tube is then slowly rotated till the joint appear in profile as two parallel lines. After cleaning and drapping and administration of local anesthesia a22-g spinal needle is inserted in line with x-ray beam till bony contact is felt. All procedures will be performed under sterile conditions. Each facet joint is infiltrated with a mixture containing 0.5 ml of 0.25 % bupivacaine and 0.5 ml (20mg) methylprednisolone acetate injected into the joint.)
  Arms: Group 1(Fluoroscopy guided group)
Procedure: Ultrsound guided Facet joint injection — Ultrsound guided Facet joint injection (Patients will be placed in a prone position. The needle is inserted 1-2 cm laterally from the midline at the lateral end of the transducer and precisely positioned in the US plane at an angle of approximately 45o with respect to the axial plane)
  Arms: Group2 (Ultrasound guided group)

SUMMARY:
The aim of this study is to compare the efficacy of fluoroscopy guided lumbar facet joint injection versus ultrasound guided injection in patients with low back pain due to facet syndrome.

DETAILED DESCRIPTION:
All patients will be randomly classified into two equal groups (40 patients each) by using closed envelops, a computer generated random allocation codes.

Group 1(Fluoroscopy guided group) (n =40 patients):

The patient will be placed in the prone position with a pillow under the abdomen to correct the lumbar lordosis. The joint to be injected is located and marked, the x ray tube is then slowly rotated till the joint appear in profile as two parallel lines. After cleaning and drapping and administration of local anesthesia a22-g spinal needle is inserted in line with x-ray beam till bony contact is felt. All procedures will be performed under sterile conditions. Each facet joint is infiltrated with a mixture containing 0.5 ml of 0.25 % bupivacaine and 0.5 ml (20mg) methylprednisolone acetate injected into the joint.

Group2 (Ultrasound guided group) (n=40 patients):

Patients will be placed in a prone position. Posterior paravertebral parasagittal sonograms will be obtained to identify of the different spinal levels. The spinous process and adjacent structures (lamina of the vertebral arch, facet joint, accessory process, and mammillary process) will be delineated by transverse sonograms at the target level, and the midpoint of the facet joint space will be established. After cleaning and drapping and administration of local anesthesia. If the joint is clearly or partially visible, a spinal needle is advanced under US guidance into the joint space of each lumbar facet joint. The needle is inserted 1-2 cm laterally from the midline at the lateral end of the transducer and precisely positioned in the US plane at an angle of approximately 45owith respect to the axial plane until the needle tip reached the target and bony contact is felt. This enables visualization of the needle, which appears as a bright line-shaped echo pattern on the transverse sonogram. If the needle placement is correct, a mixture containing 0.5 ml of 0.25 % bupivacaine and 0.5 ml(20mg) methylprednisolone acetate is administered intra-articular (until resistance was encountered) and injected around the posterior facet joint capsule.

ELIGIBILITY:
Inclusion Criteria:

* Patients, more than 18 years old, with pain associated with lumbar hyper-extension, lateral flexion, and tenderness on paravertebral regions corresponding to facet joints but normal findings on the straight leg raise test and neurologic examination.

Exclusion Criteria:

* Patient refusal and lack of consent.
* Local or systemic infection.
* allergy to steroids or local anesthetics
* Patients with coagulopathies.
* Evidence of nerve root compression at the expected level on MRI.
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Success rate of the technique | 1 day
  Success rate of the technique

SECONDARY OUTCOMES:
The visual analogue scale (VAS) score | Up to 3 months
  The visual analogue scale (VAS) score: before injections and at 1hour,a week, a month, and three months after injections.
Oswestry disability index. (ODI) | Up to 3 months
  (Pain Intensity, Personal Care, Lifting, Walking, Sitting, Standing, Sleeping, Sex Life, Social Life and Traveling )
Duration of procedure | 2 hours
  Duration of procedure
Complications | 1 week
  Allergy, infection

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Abogabal, MSc., Principal Investigator — Anesthesia, ICU and pain medicine department of Tanta university
Locations (1):
- Anesthesia , ICU, and pain medicine department, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No